CLINICAL TRIAL: NCT02118246
Title: The Clinical Effects of Dry Needling & Kinesio Tape on Myofascial Trigger Point in the Vastus Lateralis Muscle in Subjects With PFPS
Brief Title: The Effects of Dry Needling & Kinesio Tape on Anterior Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Welfare and Rehabilitation Science (Other)
Responsible Party: Principal Investigator, Amir Massoud Arab, Dr., University of Social Welfare and Rehabilitation Science
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 930127
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Knee pain,Dry Needling, kinesioTape,Trigger point
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Dry Needling; Athletic Tape

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dry Needling (Experimental): The taut band of trigger point in vastus lateralis muscle; localized between the thumb and index finger, was needled forward and backward repeatedly until there were no more local twitch response
  Interventions: Device: Dry Needling
- Kinesio Tape (Experimental): Y technique with 25% tension on the tails was applied. Direction of the technique was insertion to origin of the muscle and zone of the trigger point was placed at the center of Y strip.
  Interventions: Device: Kinesio Tape

INTERVENTIONS:
Device: Dry Needling — Dry needling was performed for one week, three times a week.
  Other Names: Western Accupuncture
  Arms: Dry Needling
Device: Kinesio Tape — Kinesio tape was performed for one week, three times a week.
  Other Names: Kenso Tape
  Arms: Kinesio Tape

SUMMARY:
Patellofemoral Pain Syndrome(PFPS) is one of the most common health-related complaints in today's societies. Myofascial pain syndrome(MPS) have been attributed as the main cause and primary source of musculoskeletal pain. Trigger point of the vastus lateralis muscle may pull the patella superiorly and laterally, increasing compression of the patellofemoral joint during physical activities, result in PFPS and anterior knee pain. The purpose of this study was to investigate the effects of Dry Needling & kinesio tape on trigger point of vastus lateralis muscle in PFPS subjects.

DETAILED DESCRIPTION:
Pain intensity, pain pressure threshold and Disability of knee were collected at base line and at the end of treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of a palpable taut band in muscle.
2. Presence of a hypersensitive tender spot in the taut band.
3. Reproduction of the typical referred pain pattern of the trigger point in response to compression. To detect active trigger point, trigger point pressure tolerance was assessed using a mechanical pressure algometer. The investigator applied continuous pressure with the algometer with an approximate pressure of 2.5 kg/cm2.
4. Spontaneous presence of the typical referred pain pattern and/or patient recognition of the referred pain as familiar.

5- Pain of at least 30 mm on a visual analogue scale (VAS) from 0 mm (no pain) to 100 mm (worst imaginable pain).

Exclusion Criteria:

1. had a history of fracture of knee joint, dislocation of patella
2. previous knee or ankle surgery
3. had a history of neurologic condition
4. having physical therapy within the past month before the study
5. pregnancy
6. taking anticoagulants (e.g. warfarin)
7. local infection

Ages: 20 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Pain | one year
  Pain intensity using Visual Analogue Scale (VAS) were collected at base line and at the end of treatment

SECONDARY OUTCOMES:
pain pressure threshold | one year
  A pressure threshold algometer was used to measure the pain pressure threshold of a Trigger point of the vastus lateralis muscle before treatment and the end of treatment(after one week).

OTHER OUTCOMES:
knee disability | one year
  The knee osteoarthritis outcome scale(KOOS) questionnaire was used to assess the knee disability.

CONTACTS AND LOCATIONS:
Overall Officials: Amir M Arab, PhD, Principal Investigator — University of Social Welfare and Rehabilitation Science
Locations (1):
- University of Social Welfare and Rehabilitation Sciences, Tehran, Islamic Republic of, Iran